CLINICAL TRIAL: NCT04490460
Title: Evaluation of the Safety and Effects on Glycemic Control of Medical Food Formulation WBF-0031 in Subjects With Abnormal Glucose Tolerance
Brief Title: Effects on Glycemic Control of WBF-0031 in Subjects With Abnormal Glucose Tolerance
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Eden Miller (Industry)
Collaborators: Pendulum Therapeutics (Industry)
Responsible Party: Sponsor-Investigator, Eden Miller, Principal Investigator, Diabetes and Obesity Care
Organization: Diabetes and Obesity Care (Industry)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: WB01-501
Record Dates: First submitted 2020-07-13; First posted 2020-07-29 (Actual); Last update posted 2020-07-29 (Actual); Status verified 2020-07

CONDITIONS: Abnormal Glucose Tolerance

STUDY DESIGN:
Intervention Model Description: Balanced randomization first arm, formulation WBF-0031 and placebo. Second arm all subjects formulation WBF-0031.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Study product was provided for each arm in identical capsules.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- First 12 Weeks (Placebo Comparator): 1 capsule administered twice daily with morning and evening meal for 12 weeks. Double blind 50% Placebo capsules identical to those containing WB-0031 and 50% WB-0031
  Interventions: Dietary Supplement: WBF-0031
- Second 12 Weeks (Active Comparator): 1 capsule administered twice daily with morning and evening meal for 12 weeks. All participants receiving WB-0031.
  Interventions: Dietary Supplement: WBF-0031

INTERVENTIONS:
Dietary Supplement: WBF-0031 — Medical food formulation WBF-0031

SUMMARY:
Evaluation of the safety and effects on glycemic control of medical food formulation WBF-0031 in subjects with abnormal glucose control.

DETAILED DESCRIPTION:
The current study aims to investigate if altering the microbiome though Pendulum Glucose Control supplementation can have implications aimed at maintaining normal blood glucose levels that are critical for preventing diabetes and its metabolic complications. The experimental design consists of two-12 week treatment periods in subjects with prediabetes, as defined by the National Diabetes Prevention Program (DPP) criteria.

The first study period of 12 weeks will be double-blinded, placebo-controlled. The Pendulum Glucose control and placebo will be in a capsule form and identical in appearance, and dispensed to each participant according to the randomization schedule in the first 12 weeks. All subjects will receive the active product (Pendulum Glucose Control) in the second, subsequent 12 week period.

Fasting total cholesterol, triglycerides, LDL, and HDL cholesterol, Fasting insulin and Glucose, High sensitivity C Reactive Protein (hsCRP), Chemistry 14, and HbA1c will be obtained at baseline, and during first and second study period, as well as vital signs of weight, BP, and waist circumference.

In addition, CGM (Abbott System Freestyle Libre Pro) data collection will be done three times during the study as noted in Schedule of Events. Baseline Blinded CGM will be performed for approximately 14 days prior to starting the intervention with Pendulum Glucose Control. Second Blinded CGM period for approximately 14 days will occur mid-way through the intervention (weeks 5 and 6) and a third period of Blinded CGM wear will occur during the last 2 weeks of the intervention (weeks 11 and 12). During the Baseline, study period one and period 2 a mixed meal tolerance consisting of 2 Boost Shakes will be given on day 5 of each sensor wear.

At the completion of the study, analysis of the vital signs, laboratory values, CGM data for average glucose, standard deviation, TIR (time in range), as well as glycemic results of MMT for each time interval; baseline, study period one, and two.

ELIGIBILITY:
Inclusion Criteria:

1. Between 18-80 years of age
2. BMI < 45 kg/m2
3. Eligible based on a recent (within the past year) blood test meeting one of these specifications:

   1. Fasting glucose of 100 to 125 mg/dl
   2. Plasma glucose measured 2 hours after a 75-gram glucose load of 140 to 199 mg/dl
   3. A1c of 5.7 to 6.4%
   4. Clinically diagnosed gestational diabetes mellitus (GDM) during a previous pregnancy (may be self-reported)
4. Willing to comply with study requirements
5. Provide written informed consent

Exclusion Criteria:

1. Known diagnosis of diabetes / taking any medication for the treatment of diabetes including the off-label use of a GLP-1 receptor agonist, SGLT-2, or metformin) within the last 3 months for weight loss.
2. Active participation in another lifestyle or behavior change education or research program (DPP or weight loss program)
3. Current treatment with systemic corticosteroids (topical and nasal steroids are allowed)
4. Subjects who have received an antibiotic, antifungal, antiparasitic, or antiviral treatment within 30 days prior to study entry
5. Pregnant women

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2020-06-01 (Actual); Primary Completion 2021-02-01 (Estimated); Study Completion 2021-02-28 (Estimated)

PRIMARY OUTCOMES:
Safety Assessment of Adverse Events | 30 weeks
  Safety assessed via spontaneous adverse events reported during the study period and changes in chemistry 14 panel
Time spent in target blood glucose | Three 14 day intervals
  Difference in daily glucose levels as measured by the amount of time spent in target blood glucose for each CGM wear period. Adjustable glucose thresholds will be set as follows:<60 mg/dL, <70 mg/dL, >140 mg/dL, >180 mg/dL and >240 mg/dL. The percent of values above, below, and between these points will be calculated.

SECONDARY OUTCOMES:
Total Glucose Area Under the Curve (AUC) from baseline | 24 weeks
  Twelve and 24 week difference from baseline in total Glucose AUC during a standard Meal Tolerance Test (MMT)
Incremental Glucose Area Under the Curve (AUC) from baseline | 24 weeks
  Twelve and 24 week difference from baseline in incremental Glucose AUC during a standard Meal Tolerance Test (MMT)
Glucose peaks | 30 weeks
  Mean and standard deviation of post-prandial peak glucose and time to peak for each meal
A1c | Week 0, Week 12, Week 24
  Improvement in A1c measured as a change in A1c levels from baseline at 12 and 24 weeks. Subjects enrolled in the study will have fasting A1c measurements at the time of enrollment and weeks, 0, 12 and 24 weeks.

OTHER OUTCOMES:
Questionnaire | Week 0, Week 12, Week 24
  Quality of life questionnaire responses measured at 0, 12 and 24 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Eden Miller, D.O., Principal Investigator — Diabetes and Obesity Care
Locations (1):
- Diabetes and Obesity Care, Bend, Oregon, United States

IPD SHARING:
Plan to Share IPD: No